CLINICAL TRIAL: NCT05465395
Title: Effects of Upper Cervical and Thoracic Chiropractic Adjustments on the Autonomic Nervous System and Perceived Stress Response
Brief Title: Upper Cervical and Thoracic Chiropractic Adjustment
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Prioritizing other studies
Sponsor: Life University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: I-0020
Record Dates: First submitted 2022-03-07; First posted 2022-07-19 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Stress
Keywords: Heart Rate Varability; Autonomic Nervious System; Chiropractic Adjustment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upper Cervical Adjustment (Experimental): Upper cervical adjustemnt
  Interventions: Procedure: Upper Cervical Adjustemnt; Procedure: Thoracic Adjustemnt
- Thoracic Adjustment (Active Comparator): Thoracic adjustment
  Interventions: Procedure: Upper Cervical Adjustemnt; Procedure: Thoracic Adjustemnt

INTERVENTIONS:
Procedure: Upper Cervical Adjustemnt — Upper cervical adjustement
Procedure: Thoracic Adjustemnt — Thoracic adjustment

SUMMARY:
The proposed study examines the differences in how the ANS responds to cervical adjustments in comparison to thoracic adjustments. This study is the continuation of a previous study titled Perceived stress and patterns of autonomic function: a protocol development study. Autonomic tests such as HRV, GSR, and the stress surveys will be the primary method of measurement. CareTaker and Biopac devices will provide continual data collection of ECG (for HRV analysis) and GSR throughout the exam and adjustment. Participant's subjective stress levels will be measured through the use of stress questionnaires including the National Stressful Events Survey Acute Stress Disorder Short Scale, the Hamilton Anxiety Rating Scale, and the Connor-Davidson Resilience Scale. The objective of the study is to determine if the location of a chiropractic adjustment will affect the autonomic nervous system in such a way that PNS or SNS activation increases or decreases after the adjustment. Further, the study will continue to examine how the chiropractic adjustment affects the subjective stress response.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 19
* In good health
* Willing to have blood pressure taken
* Willinig to shave a small area of chest hair for placement of a ECG patch
* Consent to a physical exam
* Consent ot chiropractic evaluationa nd 2 adjustments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Caretaker Heart Rate Variability | Through study completion, an average of 1 week
  HRV allows for an understanding of Autonomic (parasympathetic) function, via measuring the interval of R peaks in QRS complexes.
Galvanic Skin Response | Through study completion, an average of 1 week
  Galvanic Skin response gives a strong measure of Sympathetic response via electrical conductivity of perspiration.
Hamilton Anxiety Rating Scale | Through study completion, an average of 1 week
  Measures the severity of anxiety symptoms
NSESSS | Through study completion, an average of 1 week
  Measures PTSD symptoms in people 18 and up.
CD-RISC-25 | Through study completion, an average of 1 week
  Measure of adaptability

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Sullivan, Study Director — Life Univeristy
Locations (1):
- Dr. Sid E. Williams Center for Chiropractic Research, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No